CLINICAL TRIAL: NCT07057167
Title: Prediction of Ovarian Cancer Histotypes and Surgical Outcome Through Artificial Intelligence
Brief Title: Prediction of Ovarian Cancer Histotypes and Surgical Outcome
Acronym: PANtHer-AI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7504
Record Dates: First submitted 2025-06-27; First posted 2025-07-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Metastatic Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic Laparoscopy videos — Diagnostic laparoscopy videos will be collected and stored on internal hard drives.
  Pseudo-anonymized laparoscopic videos will be annotated by expert clinicians. Artificial intelligence (AI)-based solutions will be developed, trained, and validated.

SUMMARY:
The standard treatment for advanced ovarian cancer (AOC) is primary cytoreductive surgery (PCS) followed by adjuvant chemotherapy. However, optimal cytoreduction is not always achievable, particularly in cases with high tumor burden or patient frailty. In such scenarios, neoadjuvant chemotherapy (NACT) followed by interval cytoreductive surgery (ICS) represents a valid alternative with comparable oncologic outcomes in selected patients.

To optimize surgical strategy, objective tools are needed to identify the best candidates for PCS. Scoring systems such as the Fagotti Score and the Predictive Index Value (PIV) assess tumor resectability, but their accuracy largely depends on surgeon expertise.

It has already developed the PREDAtOOR project, a significant advancement in the use of artificial intelligence (AI) for managing AOC. PREDAtOOR has demonstrated high accuracy in both predicting the Fagotti Score and segmenting lesions from diagnostic laparoscopy videos, thus supporting a more objective and reproducible surgical decision-making process.

Importantly, therapeutic strategies should also consider tumor biology, as the response to NACT varies across histological and molecular subtypes. Unfortunately, such information is usually derived from histopathological and genomic analyses performed only after the surgical decision.

Kurman and Shih proposed a dualistic model of epithelial ovarian tumors, with distinct clinical and molecular features:

Type I tumors (low-grade serous, endometrioid, clear cell, mucinous): indolent growth, typically confined to the ovary, with stable genomes. Early-stage cases may be cured surgically. Metastatic Type I tumors tend to be chemoresistant but may respond to targeted therapies.

Type II tumors (high-grade serous carcinoma [HGSC], carcinosarcomas, undifferentiated carcinomas): aggressive behavior, marked genomic instability, and frequent homologous recombination deficiency (HRD). Although initially sensitive to platinum-based chemotherapy and PARP inhibitors, resistance often emerges.

Among these, HGSC is the most frequent and lethal. Yet, even within HGSC, substantial variability in chemotherapy response and clinical outcome is observed. A recent morphologic classification of HGSC stratifies tumors into infiltrative vs. expansive patterns, associated with specific molecular alterations and therapeutic responses.

However, these morphological and molecular features are not yet integrated into intraoperative decision-making, highlighting a need for new intraoperative tools to personalize care.

In this precision medicine landscape, AI, particularly through machine learning and computer vision, offers powerful solutions. These technologies can process large, heterogeneous datasets and automate intraoperative assessments, enhancing objectivity and diagnostic reproducibility. While AI-based classification of histologic and molecular subtypes from laparoscopy remains largely unexplored, it holds the potential to revolutionize treatment stratification in AOC.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years of age
* Patients fit for upfront cytoreductive surgery.
* Patients undergoing diagnostic laparoscopy as part of the upfront decision-making algorithm.
* Patients with a primary diagnosis of advanced ovarian carcinoma, FIGO stage IIIB - IVB
* Signature of the informed consent / consent for the processing of personal data and associated data for research purposes in patients treated at the Fondazione Policlinico Universitario A. Gemelli IRCCS (form 743 or form pro.1145.001) / substitute declaration for the consent form for deceased patients.

Exclusion criteria:

* Lack of information on surgical outcome and clinical-pathological characteristics.
* Ovarian carcinoma patients without evidence of macroscopic peritoneal carcinomatosis (FIGO stage I-IIIA).
* Secondary cytoreductive surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced ovarian cancer who underwent diagnostic laparoscopy at the time of diagnosis, with or without subsequent cytoreductive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Computer Vision Algorithm in Predicting Ovarian Cancer Histotype | 36 months
  Proportion (%) of laparoscopic videos in which the computer vision algorithm correctly predicts the histotype of ovarian cancer (Non-Epithelial vs Epithelial, and Epithelial subtypes: Type I vs Type II), using final histopathological diagnosis as the reference standard.

SECONDARY OUTCOMES:
Accuracy of Computer Vision Algorithm in Predicting Morphological Classification | 36 months
  Proportion (%) of laparoscopic videos of high-grade serous ovarian cancer (HGSOC) in which the computer vision algorithm correctly classifies the tumor into two distinct morphological subtypes (as defined by Handley et al.) during diagnostic laparoscopy, using expert pathological assessment as the reference standard.
Accuracy of Computer Vision Algorithm in Predicting Molecular and Genetic Tumor Profiles | 36 months
  Proportion (%) of laparoscopic videos in which the computer vision algorithm correctly predicts molecular and genetic tumor profiles (homologous recombination deficiency [HRD] status, homologous recombination proficiency [HRP] status, and BRCA mutation status) using molecular/genetic testing as the reference standard.
Accuracy of Computer Vision Algorithm in Predicting Chemosensitivity or Chemoresistance in High-Grade Serous Ovarian Cancer (HGSOC) | 36 months
  Proportion (%) of laparoscopic videos of high-grade serous ovarian cancer (HGSOC) in which the computer vision algorithm correctly predicts chemosensitivity (platinum-free interval [PFI] > 6 months) or chemoresistance (PFI < 6 months), using clinical follow-up as the reference standard.
Accuracy of Computer Vision Algorithm in Predicting the Feasibility of Achieving Complete Gross Resection (CGR) | 36 months
  Proportion (%) of laparoscopic videos in which the computer vision algorithm correctly predicts the feasibility of achieving complete gross resection (CGR; defined as no visible residual disease at the end of surgery), compared with the actual surgical outcome documented by surgical reports

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fagotti, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS